CLINICAL TRIAL: NCT05344469
Title: A Non-interventional Study Evaluating Injectable Treatments (Ofatumumab, Glatiramer Acetate and Interferon β1) in Patients With Relapsing Multiple Sclerosis [AIOLOS]
Brief Title: A NIS Evaluating Injectable Treatments in Patients With Relapsing Multiple Sclerosis
Acronym: AIOLOS
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GDE02
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; RMS; NIS; ofatumumab
MeSH Terms: interventions — ofatumumab; Glatiramer Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Ofatumumab: Patients treated with ofatumumab
  Interventions: Other: ofatumumab
- Standard of Care (SoC): Patients treated with either interferon β1 (IFN-β1) or glatiramer acetate (GA)
  Interventions: Other: glatiramer acetate; Other: interferon β1

INTERVENTIONS:
Other: ofatumumab — There is no treatment allocation. Patients administered ofatumumab by prescription that have started as routine medical treatment will be enrolled.
  Groups: Ofatumumab
Other: glatiramer acetate — There is no treatment allocation. Patients administered glatiramer acetate by prescription that have started as routine medical treatment will be enrolled.
  Groups: Standard of Care (SoC)
Other: interferon β1 — There is no treatment allocation. Patients administered interferon β1 by prescription that have started as routine medical treatment will be enrolled.
  Groups: Standard of Care (SoC)

SUMMARY:
This is an observational, non-interventional, multicenter, open-label study in patients being treated with any approved injectable Disease-modifying Therapy (DMT) for Relapsing Multiple Sclerosis in Germany. Prospective, primary data will be collected via questionnaires and an electronic case report form (eCRF) over a period of up to approx. two years of treatment. Additionally, medical history of participants will be collected including disease duration, EDSS, MRI parameters and relapses.

DETAILED DESCRIPTION:
The prerequisite for participation in this observational study is the independent decision of the treating physician and patient to start an approved injectable DMT for RMS as routine medical treatment. This decision must have been made prior to enrollment in this study.

The prospective observational period per patient will be up to approx. two years from the time of consent (2 years +2 months visit window). The observational period will not be dictated by the protocol. The follow-up documentation will take place at a frequency defined as per investigator's discretion. The diagnostic or monitoring procedures are only those ordinarily applied to the therapeutic strategy and to routine clinical care, can be performed as telemedicine visits and will take place as per investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Male or female patients aged ≥18 years at enrollment
3. Diagnosis of MS according to the 2017 revised McDonald criteria (Thompson et al 2018b)
4. RMS with active disease as defined by Lublin et al. (2014)
5. Max. 1 relapse during the previous year and max. 2 relapses during the previous two years prior to enrollment
6. Disability status at enrollment with an EDSS score of 0 to 2.5 (inclusive)
7. Planned initiation or initiation within the past 14 days with an approved injectable DMT for MS as routine medical treatment

Exclusion Criteria:

1. Patients being treated outside of the approved label
2. > 5 years since first symptom(s) (leading to MS diagnosis) at enrollment
3. Previous therapy with any DMT for the treatment of MS prior to enrollment (except within the past 14 days with an approved injectable DMT for MS as routine medical treatment; see Inclusion criteria #7)
4. Relapse prior to enrollment which has led to a severe deficit relevant to everyday life upon discretion of the investigator after exhaustion of the relapse therapy
5. Poor recovery from the first two relapses prior to enrollment upon discretion of the investigator
6. EDSS Functional System Score "Pyramidal Functions" ≥ 2 at enrollment
7. Simultaneous participation in any investigational trial or simultaneous participation in another Novartis-sponsored non-interventional study with Ofatumumab

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with planned initiation or initiation within the past 14 days with an approved injectable DMT for RMS as routine medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who continue to receive their first-line treatment | Month 24
  Proportion of patients who continue to receive their first-line treatment (ofatumumab or injectable SOC therapies (IFN-β1 or GA))

SECONDARY OUTCOMES:
Proportion of patients who continue to receive their first-line treatment | Month 12
  Proportion of patients who continue to receive their first-line treatment (ofatumumab or injectable SOC therapies (IFN-β1 or GA))
Impact of first-line treatment on health economy | Baseline, month 6, month 12, month 18 and month 24
  Mean annual health care resource utilization cost, annual direct medical costs, annual direct nonmedical costs and annual indirect costs as measured by MS Health Resource Utilization Survey [MS-HRS]
  MS-HRS is a 24-item questionnaire covers societal resource use, regardless of the issue of reimbursement, as well as impact of the disease on work, family and leisure. With the help of this questionnaire a monetary value can be assigned to e.g. the stage of MS, a relapse or a therapy.
Fatigue Symptoms and Impact Questionnaire-RMS | Baseline, month 3, month 6, month 12, month 18, month 24
  Fatigue Symptoms and Impact Questionnaire-RMS [FSIQ-RMS]
  The FSIQ-RMS comprises 20 items organized in a conceptual framework with 2 symptom domains (energy, muscle weakness) and 7 impact domains (daily activities, cognition, emotions, physical impact, self-care, sleep, social impact) in order to measure fatigue symptoms and impacts in relapsing multiple sclerosis.
  A scoring algorithm standardizes scores on both the symptoms domain (daily and weekly) and impacts subdomains (weekly) to a 0 to 100 scale, with higher scores indicating more severe symptoms and impacts. There is no single summary score across the FSIQ-RMS instrument, but rather 1 symptoms score and 3 impacts subdomain scores.
Patient Health Questionnaire 8 [PHQ-8] | Baseline, month 3, month 6, month 12, month 18, month 24
  The PHQ-8 is a valid diagnostic and severity measure for depressive disorders. It consists of eight items, each of which is scored 0 to 3, providing a 0 to 24 severity score. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Generalized Anxiety Disorder Scale 7 [GAD-7] | Baseline, month 3, month 6, month 12, month 18, month 24
  The GAD-7 is a validated 7-item anxiety scale to diagnose generalized anxiety disorder. Each of the items is scored 0 to 3, providing a 0 to 21 severity score. Scores of 5, 10, and 15 represent cutpoints for mild, moderate, and severe anxiety, respectively
MS Treatment Concerns Questionnaire [MSTCQ] | Baseline, month 3, month 6, month 12, month 18, month 24
  MS Treatment Concerns Questionnaire [MSTCQ] is used to assess participants' satisfaction with their treatment injections.
  The MSTCQ includes 20 items pertaining satisfaction with the injection system (including issues related to use of the device and preparation of the medication for injection), and AEs related to the patient MS treatment.
  All questions have a 5-point response choice, with the responses scored between 1-5. The MSTCQ scores are formed as the sum of all scores. The maximum total score is 100. Lower scores indicate a better state.
Expanded disability status scale (EDSS) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  EDSS is a widely used and accepted instrument to evaluate disability status at a given time and, longitudinally, to assess accumulation of disability in clinical studies in MS. The EDSS scale consists of scores in each of seven functional systems (FSs) and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The FSs are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions (Fatigue contributes)
Time to onset of confirmed disability progression (CDP) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Time to onset of confirmed disability progression (CDP) defined as an increase from baseline in EDSS sustained for at least 3 and 6 months, respectively
Proportion of patients with confirmed disability progression (CDP) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Proportion of patients with confirmed disability progression (CDP) defined as an increase from baseline in EDSS sustained for at least 3 and 6 months, respectively
Time to onset of confirmed disability improvement (CDI) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Time to onset of confirmed disability improvement (CDI) defined as a decrease from baseline in EDSS sustained for at least 3 and 6 months
Proportion of patients with CDI | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Proportion of patients with CDI defined as a decrease from baseline in EDSS sustained for at least 3 and 6 months
T1 Gd-enhancing lesions per brain | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  T1 Gd-enhancing lesions per brain to be measured
Annualized T2 lesion rate | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  New or enlarging T2 lesions per brain and per year (annualized T2 lesion rate)
Proportion of patients with no evidence of disease activity (NEDA3) upon discretion of the investigator. | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Proportion of patients with no evidence of disease activity (NEDA3) upon discretion of the investigator. NEDA3 is defined as no 3mCDP, no confirmed MS relapse and no new or enlarging T2 lesions on any MRI scan compared to baseline
Proportion of patients with no clinical disease activity and no discontinuation of current treatment due to AEs | Up to 24 months
  Proportion of patients with no clinical disease activity measured by relapse and disease progression and no discontinuation of current treatment due to AEs (excluding pregnancies) and lack of effectiveness
Annualized relapse rate | Up to 24 months
  Annualized relapse rate, defined as the number of confirmed Multiple Sclerosis relapses in a year.
  Relapse defined as an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must have been present for at least 24 hours and occurred in the absence of fever (< 37.5°C) or a known infection.
Time to first relapse | Up to 24 months
  Relapse defined as an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must have been present for at least 24 hours and occurred in the absence of fever (< 37.5°C) or a known infection.
Proportion of relapse free patients | Up to 24 months
  Relapse defined as an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must have been present for at least 24 hours and occurred in the absence of fever (< 37.5°C) or a known infection.
Number of patients and reasons for discontinuation of treatment | Up to 24 months
  Number of patients and reasons for discontinuation of treatment classified by category:
  * efficacy (e.g. occurrence of relapse, evidence of disease activity in MRI)
  * safety and tolerability (e.g. injection-site reactions, influenza-like symptoms)
  * or convenience (e.g. inconvenient administration, frequency of injections)
Proportion of patients who continue to receive their subsequent treatment | Up to 24 months
  Proportion of patients who, at a given time over the period of 2 years, continue to receive their subsequent treatment
Reasons for and number of treatment interruptions per patient | Up to 24 months
  Reasons for and number of treatment interruptions per patient to be collected
Duration of treatment interruptions per patient | Up to 24 months
  Duration of treatment interruptions per patient to be collected
Number of patients with treatment interruptions | Up to 24 months
  Number of patients with treatment interruptions to be collected
Proportion of drug-related adverse events (AEs) | Up to 24 months
  Proportion of drug-related adverse events (AEs) including those of special interest (main focus on injection site reactions such as scarring, skin reactions)
Persistence of drug-related adverse events (AEs) | Up to 24 months
  Persistence of drug-related adverse events (AEs) including those of special interest (main focus on injection site reactions such as scarring, skin reactions, influenza-like symptoms)
Specific safety assessment of injection related AEs | Up to 24 months
  Specific safety assessment of injection related AEs. (i.e. injection site reaction AEs vs. injection systemic reaction AEs) summarized by providing the number and percentage of patients with each of the symptoms and pre-specified grouping of symptoms as well as overall.
Proportion of participants discontinuing treatment due to insufficient effectiveness (lack of efficacy) or tolerability/safety reasons | Up to 24 months
  Proportion of participants discontinuing treatment due to insufficient effectiveness (lack of efficacy) or tolerability/safety reasons
Presence of spinal cord lesions | Baseline, month 3,month 6, month 9, month 12, month 15, month 18, month 21, month24
  Proportion of patients with spinal cord lesions present

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- Germany (72):
  - Novartis Investigative Site, Hettingen, Baden-Wurttemberg
  - Novartis Investigative Site, Schwaebisch, Baden-Wurttemberg
  - Novartis Investigative Site, Schwetzingen, Baden-Wurttemberg
  - Novartis Investigative Site, Bamberg, Bavaria
  - Novartis Investigative Site, Untermeiting, Bavaria
  - Novartis Investigative Site, Bad Homburg, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Wildeshausen, Lower Saxony
  - Novartis Investigative Site, Meerbusch, North Rhine-Westfalia
  - Novartis Investigative Site, Altenburg
  - Novartis Investigative Site, Altenholz
  - Novartis Investigative Site, Alzey
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Bergneustadt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Gladenbach
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lünen
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mettmann
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Montabaur
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nagold
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Saalouis
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Weil der Stadt

IPD SHARING:
Plan to Share IPD: No